CLINICAL TRIAL: NCT01193751
Title: Prospective Multicenter Study to Evaluate the Validity of the Specified Apgar-score in Asphyxiated Infants Under Resuscitation
Brief Title: Apgar-Score in Asphyxiated Infants Under Resuscitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Prof. Dr. Mario Rüdiger, Dresden University of Technology, Department of Neonatology
Other Study IDs: Apgar in asphyxiated infants
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2010-09

CONDITIONS: Death; Neurodevelopmental Impairment
Keywords: Birth Asphyxia; Newborn's Resuscitation; Death; Neurodevelopmental Impairment
MeSH Terms: conditions — Death; Asphyxia Neonatorum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- asphyxiated newborns > 37 weeks of gestation

SUMMARY:
The specified Apgar-Score in combination with the AAP-Score predicts the morbidity and mortality of asphyxiated newborns.

DETAILED DESCRIPTION:
In the first place the Apgar-score helps to evaluate the postnatal adaptation of the newborn and is used as an index for resuscitative interventions. However, it has been shown in the past that the score has its limits and may be influenced by several factors such as the variability of the examiner, drugs, parental age, neurological impairment of the child as well as premature delivery. Previous studies have proven, however, that the evaluation of the infant's condition with the conventional Apgar-score is affected due to non-uniform definitions.

For this, an explanation might be that on the one hand the inaccuracy of the score is based on missing guidelines for the assessment of the score in premature infants. Both, muscle tone and reflexes of extremely premature infants are physiologically more immature than they are in term newborns. In conclusion, healthy premature infants often achieve a lower Apgar-score than their term counterparts. However, this is rather an expression of their immaturity than a sign for postnatal depression.

Another reason for the inaccuracy of the score might have its origin in the limited comparability and validity of the Apgar-score when applied in resuscitated newborns. Until now there is no consensus how to assess the condition of the newborn under resuscitation, since the individual characteristics composing the score are affected by the resuscitation itself. For example, heart frequency and skin colour are improved by sufficient ventilation. So far there are no regulations on how this fact should be considered while assessing the score. A description of the infant's condition without interventions respectively with interruption of the interventions applied would be in contrast to Apgar's intention to have a score "which could be determined easily without interfering with the care of the infant". The description of the condition independently of the interventions applied offers a practicable alternative. By using this method the resuscitation will not be interrupted and the score will not express the efforts of the infant but describe its condition, independently of the requirements needed to achieve this condition.

To validate the accuracy of the specified version of the Apgar-score to predict neonatal mortality and long term outcome in preterm infants, the multicenter TEST-Apgar study has been performed recently.

The American Academy of Pediatrics (AAP) is also aware of the problem concerning the description of resuscitated newborns. As a solution, it was suggested to use an expanded Apgar-score reporting form that accounts for concurrent resuscitative interventions (AAP-Score). This way the infant's condition can be estimated and documented more easily. Although the AAP-Score has been suggested 4 years ago, data on the predictive reliability are not available yet. This aspect regarding the neonatal mortality of premature infants has also been analyzed in the TEST-Apgar study. The results show that the specified Apgar-Score should be used in combination with the AAP-Score in the future to appraise the condition of premature infants. Its predictive value regarding the neonatal mortality of premature infants is very good. Detailed results will be published soon.

The present study analyzes the validity of the specified Apgar- and the AAP- Scores in asphyxiated infants >37 weeks of gestation undergoing resuscitation. Since the Apgar-score presents an index for the postnatal adaption to the extra-uterine life, reflects the efficiency of resuscitative interventions and also serves as an inclusion criteria for specific types of therapy (e.g. hypothermia therapy), it is necessary, to standardise the use of the Apgar-score and improve its prognostic value.

ELIGIBILITY:
Inclusion Criteria:

* Parental consent
* Born within the study center (inborn)
* gestational age >37 completed weeks
* Receiving one or more resuscitive intervention (CPAP, Oxygen supplementation, Intubation and ventilation, bag and mask ventilation, surfactant, catecholamines, chest compression) and/or Birth Asphyxia with a umbilical artery pH <7,0 or BE > -16 with subsequent admission to NICU.

Exclusion Criteria:

missing parental consent

Min Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Asphyxiated newborns >37 weeks of gestation receiving resuscitative interventions
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Death or Neurologic impairment | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Dresden University of Technology, Department of Neonatology, Dresden, Germany